CLINICAL TRIAL: NCT00603759
Title: the Role of COX-2 Inhibitor(CELECOXIB) in Combination With Chemoradiation in Locally Advanced Head & Neck Carcinoma, Phase III Randomized Clinical Trial
Brief Title: COX-2 Inhibitor With Concurrent Chemoradiation in Locally Advanced Head & Neck Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: department of radiation oncology (Ambiguous)
Responsible Party: Dr mahdi Aghili, department of radiation and oncology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3058
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Head and Neck Cancer
Keywords: COX2 inhibitor; head and neck cancer; chemoradiation
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: celecoxib
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: celecoxib — 100 mg qid
  Arms: 1
Drug: placebo — 1 cap qid
  Arms: 2

SUMMARY:
chemotherapy- and radiotherapy-induced oral mucositis represents a therapeutic challenge frequently encountered in cancer patients.This side effect causes significant morbidity and may delay or interrupt the treatment plan, as well reduce therapeutic index. cyclo-oxygenase 2 (COX-2) is an inducible enzyme primarily expressed in inflamed tissues and tumor. COX-2 inhibitors have shown promise as radio- and chemosensitizer and reduce radio-induced toxicities.

we have conducted a phase III, randomized double blind clinical trial to evaluate the toxicity and efficacy of celecoxib, a selective COX-2 inhibitor, administered concurrently with chemotherapy, and radiation for locally advanced head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* stage III/IV (locally advanced) carcinoma of oropharynx, oral cavity, hypopharynx, larynx, or nasopharynx
* primary treatment with chemoradiation

Exclusion Criteria:

* distant metastasis
* incomplete treatment
* adjuvant chemoradiation after surgery without apparent tumor

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2006-04; Primary Completion 2007-08 (Actual); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
efficacy of celecoxib (response rate and local control) | 30 months

SECONDARY OUTCOMES:
toxicity of celecoxib | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Mahdi Aghili, MD, Study Chair — cancer institute center
Locations (1):
- Department of Chemoradiation, Tehran, Tehran Province, Iran